CLINICAL TRIAL: NCT06310551
Title: A Phase 1 Double-Blind (Sponsor-unblinded), Placebo-Controlled Randomized, Single Ascending Dose and Multiple Dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Parenterally Administered VH4524184 in Healthy Adults
Brief Title: First Time in Human Study of Long Acting VH4524184 Formulations
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 218804
Record Dates: First submitted 2024-03-05; First posted 2024-03-15 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: HIV Infections
Keywords: Safety; Tolerability; Parenteral; First Time in Human; Pharmacokinetics; Ascending Dose; Multiple Dose; Healthy Adults
MeSH Terms: conditions — HIV Infections | interventions — hyaluronidase PH-20

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Formulation A SC Group (Experimental): Participants receive a Formulation A starting dose of VH4524184 LAI subcutaneously (SC).
  Interventions: Drug: Oral VH4524184; Drug: VH4524184 Formulation A SC; Drug: Placebo Formulation A SC; Drug: rHuPH20
- Formulation B SC Group (Experimental): Participants receive a Formulation B starting dose of VH4524184 LAI subcutaneously.
  Interventions: Drug: Oral VH4524184; Drug: rHuPH20; Drug: VH4524184 Formulation B SC; Drug: Placebo Formulation B SC
- Formulation C SC Group (Experimental): Participants receive a Formulation C starting dose of VH4524184 LAI subcutaneously. This intervention is optional and initiated only if Formulation B is poorly tolerated.
  Interventions: Drug: Oral VH4524184; Drug: rHuPH20; Drug: VH4524184 Formulation C SC; Drug: Placebo Formulation C SC
- Formulation A IM Group (Experimental): Participants receive a Formulation A starting dose of VH4524184 LAI intramuscularly (IM).
  Interventions: Drug: Oral VH4524184; Drug: VH4524184 Formulation A IM; Drug: Placebo Formulation A IM
- Formulation B IM Group (Experimental): Participants receive a Formulation B starting dose of VH4524184 LAI intramuscularly (IM).
  Interventions: Drug: Oral VH4524184; Drug: VH4524184 Formulation B IM; Drug: Placebo Formulation B IM
- Multiple doses Group (Experimental): VH4524184 LAI formulations administered SC or IM as single doses that achieve adequate PK exposure targets, may be evaluated for safety and tolerability as multiple doses.
  Interventions: Drug: Oral VH4524184; Drug: VH4524184 Formulation A SC; Drug: Placebo Formulation A SC; Drug: rHuPH20; Drug: VH4524184 Formulation B SC; Drug: Placebo Formulation B SC; Drug: VH4524184 Formulation C SC; Drug: Placebo Formulation C SC; Drug: VH4524184 Formulation A IM; Drug: Placebo Formulation A IM; Drug: VH4524184 Formulation B IM; Drug: Placebo Formulation B IM

INTERVENTIONS:
Drug: Oral VH4524184 — VH4524184 to be taken orally.
Drug: VH4524184 Formulation A SC — Low (<1mL) starting dose of VH4524184 LAI Formulation A administered subcutaneously.
  Arms: Formulation A SC Group; Multiple doses Group
Drug: Placebo Formulation A SC — Starting dose of Placebo Formulation A administered subcutaneously.
  Arms: Formulation A SC Group; Multiple doses Group
Drug: rHuPH20 — Dose of rHuPH20 administered subcutaneously.
  Other Names: PH20, Halozyme ENHANZE
  Arms: Formulation A SC Group; Formulation B SC Group; Formulation C SC Group; Multiple doses Group
Drug: VH4524184 Formulation B SC — Starting dose of VH4524184 LAI Formulation B administered subcutaneously.
  Arms: Formulation B SC Group; Multiple doses Group
Drug: Placebo Formulation B SC — Starting dose of Placebo Formulation B administered subcutaneously.
  Arms: Formulation B SC Group; Multiple doses Group
Drug: VH4524184 Formulation C SC — Starting dose of VH4524184 LAI Formulation C administered subcutaneously.
  Arms: Formulation C SC Group; Multiple doses Group
Drug: Placebo Formulation C SC — Dose of Placebo Formulation C administered subcutaneously.
  Arms: Formulation C SC Group; Multiple doses Group
Drug: VH4524184 Formulation A IM — Starting dose VH4524184 LAI Formulation A administered intramuscularly.
  Arms: Formulation A IM Group; Multiple doses Group
Drug: Placebo Formulation A IM — Dose of Placebo Formulation A administered intramuscularly.
  Arms: Formulation A IM Group; Multiple doses Group
Drug: VH4524184 Formulation B IM — Starting dose VH4524184 LAI Formulation B administered intramuscularly.
  Arms: Formulation B IM Group; Multiple doses Group
Drug: Placebo Formulation B IM — Dose of Placebo Formulation B administered intramuscularly.
  Arms: Formulation B IM Group; Multiple doses Group

SUMMARY:
The purpose of this study is to identify 1 or more doses of parenterally administered VH4524184 that are safe, well tolerated and yield a PK drug exposure profile necessary to deliver a long-acting antiretroviral therapy for the treatment of HIV-1 infection.

ELIGIBILITY:
Inclusion Criteria:

Age

1. Participant must be 18 to 55 years of age inclusive, at the time of signing the informed consent.

   Type of Participant and Characteristics
2. Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
3. Participants who are negative for SARS-CoV-2, performed on admission/readmission to the Phase 1 unit, using an approved molecular test (PCR).
4. Participants who are able to understand and comply with protocol requirements and timetables, instructions, and protocol-stated restrictions.

   Weight
5. Body weight ≥50.0 kg (110 lbs) for men and ≥45.0 kg (99 lbs) for women and body mass index within the range 18.5 to 32.0 kg/m2 (inclusive).

   Sex and Contraceptive/Barrier Requirements
6. Male or female

   1. Male Participants: No restrictions for male participants
   2. Participants of female sex assigned at birth is eligible to participate as long as the participant is not breastfeeding and is of non-childbearing potential.

   Informed Consent
7. Capable of providing signed informed consent.

Exclusion Criteria:

Medical Conditions

1. History or presence of clinical condition or disorder that could be capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study drug, interfering with the interpretation of data or would make the participant unsuitable for the study; unable to comply with dosing requirements; or unable to comply with study visits.
2. Abnormal blood pressure as determined by the investigator.
3. Lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
4. Breast cancer within the past 10 years.
5. Current or chronic history of liver disease or known hepatic or biliary abnormalities.
6. Medical history of cardiac arrhythmias or cardiac disease or a family and personal history of long QT syndrome.
7. Underlying skin disease or disorder that would interfere with the administration of study product and/or assessment of injection site reactions.
8. History of drug hypersensitivity, delayed-type hypersensitivity or severe hypersensitivity reactions, as well as history of /sensitivity to any of the study interventions including hyaluronidases.
9. Current or anticipated need for chronic anti-coagulation except for the use of low dose acetylsalicylic acid (≤325 mg) or hereditary coagulation and platelet disorders such as hemophilia or Von Willebrand Disease.
10. History of seizure.
11. Any known or suspected pre-existing psychiatric condition, including depression, anxiety and insomnia/sleep disturbances, at the discretion of the investigator.
12. Any positive (abnormal) response confirmed by the investigator or clinician (or qualified designee) administered C-SSRS at screening.
13. Insufficient muscle mass (gluteus medius or thigh) to support IM dose administration in the opinion of the investigator.
14. Presence of tattoos or skin piercings that may interfere with the administration of study product and/or assessment of ISRs, if they occur.
15. History of or on-going high-risk behaviors that may put the participant at increased risk for HIV acquisition in the opinion of the investigator. This includes participants in HIV discordant relationships, or men who report current or prior unprotected anal sex with other men and those reporting prior or current injecting drug use.

    Prior/Concomitant Therapy
16. Past or intended use of over-the-counter or prescription medication within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to dosing and for the duration of the study.
17. Receipt of any live vaccine(s) or vaccines against SARS-CoV-2 within 28 days prior to screening or 14 days before or after scheduled SC or IM dosing.

    Prior/Concurrent Clinical Study Experience
18. Exposure to more than 4 new investigational products (including long-acting investigational products) within 12 months prior to the first dosing day.
19. Current enrollment or past participation in another investigational study in which an investigational intervention was administered within the last 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product before signing of consent (OR screening) any other clinical study.
20. Participation in the study would result in loss of blood in excess of 500 mL over a 56-day period.
21. Current enrollment or past participation in this clinical study or prior participation in study 218803.

    Diagnostic Assessments
22. eGFR <60 mL/min or serum creatinine >1.1 x ULN.
23. Hemoglobin <12.5 g/dL for men and <11 g/dL for women
24. ALT or AST >1.5x upper limit of normal (ULN)
25. Total bilirubin >1.5xULN.
26. Any significant arrhythmia or ECG finding.
27. Exclusion criteria for Screening ECG - a single repeat is allowed for eligibility determination.
28. Presence of HBsAg at screening.
29. Positive Hepatitis C antibody test result at screening.
30. Positive pre-study drug/alcohol screen.
31. Positive HIV antibody test. Other Exclusions
32. Regular alcohol consumption within 6 months prior to the study defined as: An average weekly intake of >14 units for males or >7 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.
33. Regular use of known drugs of abuse.
34. Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening and at admission.
35. Sensitivity to the study drug, or components thereof, or other drug or other allergy that, in the opinion of the investigator or Sponsor Medical Monitor, contraindicates participation in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2028-01-21 (Estimated); Study Completion 2028-01-21 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants reporting adverse events (AEs) and related AEs | From first study dose administration (Day 1) up to study end (Week 52 post last dose)
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. Related AE = AE assessed by the investigator as related to the study drug.
Percentage of participants with AEs by severity | From first dose administration (Day 1) up to study end (Week 52 post last dose)
  Severity of AEs will be assessed using Division of AIDS Table for Grading the Severity of Adult Adverse Events (DAIDS). DAIDS grading scale is used to grade the toxicity associated with injection site reactions (ISR) including injection site pain (or tenderness), erythema (or redness), induration (or swelling), and pruritis. The toxicity level is graded from Grade 1 (lowest toxicity) to 4 (highest toxicity). Higher grade indicates higher toxicity.
Percentage of participants discontinuing the treatment due to AEs | From first dose administration (Day 1) up to study end (Week 52 post last dose)
Change from baseline in alanine aminotransferase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase parameters | From first dose administration (Day 1) up to study end (Week 52 post last dose)
  The liver panel laboratory parameters are assessed after the administration of long-acting injectable (LAI) VH4524184.
Change from baseline in total bilirubin parameters | From first dose administration (Day 1) up to study end (Week 52 post last dose)
  The liver panel laboratory parameters are assessed after the administration of LAI VH4524184.
Change from baseline in international normalized ratio (INR) parameters | From first dose administration (Day 1) up to study end (Week 52 post last dose)
  The liver panel laboratory parameters are assessed after the administration of LAI VH4524184.
Maximum toxicity grade increase from baseline in ALT, AST and alkaline phosphatase | From first dose administration (Day 1) up to study end (Week 52 post last dose)
Maximum toxicity grade increase from baseline in total bilirubin | From first dose administration (Day 1) up to study end (Week 52 post last dose)
Maximum toxicity grade increase from baseline in INR | From first dose administration (Day 1) up to study end (Week 52 post last dose)
Percentage of participants reporting injection site reaction (ISR) AEs | From first dose administration (Day 1) up to study end (Week 52 post last dose)
  Assessed ISRs are pain, tenderness, infections, erythema, swelling, induration, or nodules (granulomas or cysts). Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, and Grade 4 = potentially life threatening.
Duration of injection site reaction AEs | From first dose administration (Day 1) up to study end (Week 52 post last dose)
Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinity time (AUC[0-inf]) of LAI VH4524184 following single dose administration | From first dose administration (Day 1) up to study end (Week 52 post last dose)
Area under the plasma drug concentration-time curve from zero (pre-dose) to the end of the dosing interval at steady state (AUC[0-t]) of LAI VH4524184 following multiple dose administration | From first dose administration (Day 1) up to study end (Week 52 post last dose)
Maximum observed plasma drug concentration (Cmax) of LAI VH4524184 following single dose administration | From first dose administration (Day 1) up to study end (Week 52 post last dose)
Cmax of LAI VH4524184 following multiple dose administration | From first dose administration (Day 1) up to study end (Week 52 post last dose)
Time to maximum observed plasma drug concentration (Tmax) of LAI VH4524184 following single dose administration | From first dose administration (Day 1) up to study end (Week 52 post last dose)
Tmax of LAI VH4524184 following multiple dose administration | From first dose administration (Day 1) up to study end (Week 52 post last dose)
Apparent terminal half-life (t1/2) of LAI VH4524184 following single dose administration | From first dose administration (Day 1) up to study end (Week 52 post last dose)
t1/2 of LAI VH4524184 following multiple dose administration | From first dose administration (Day 1) up to study end (Week 52 post last dose)

SECONDARY OUTCOMES:
Percentage of participants with treatment emergent Grade 3 or Grade 4 laboratory abnormalities | From first dose administration of VH4524184 (Day 1) up to study end (Week 52 post last dose)
  Grade 3 is defined as causing an inability to perform usual social & functional activities with intervention or hospitalization indicated. Grade 4 is defined as an abnormality that is potentially life-threatening, causing an inability to perform basic self-care functions with intervention indicated to prevent permanent impairment, persistent disability, or death.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/